CLINICAL TRIAL: NCT06520722
Title: A New POP(Pelvic Organ Prolapse) Scoring System: Validity and Reliability
Brief Title: A New POP (Pelvic Organ Prolapse) Scoring System: Validity and Reliability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElHarty, Lecturer, Cairo University
Other Study IDs: MD-16_2023
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse; Prolapse; Prolapse, Vaginal; Prolapse Uterus; Prolapse; Cervix
Keywords: Prolapse; Pelvic organ prolapse; POP-Q; Procidentia; Uterine prolapse; Vaginal prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prolapse scoring system — A FIXED APCD classification system :
  A: Associated symptoms:
  FIXED:
  F: frequency I: infection X: sex problems E: everted mass(external protrusion of mass from the valva as PV lump sensation ,heaviness,itching and ulceration) D: digitation(patient need to digitate to complete the act of micturation or defecation)
  APCD:
  A: Dependent point on anterior wall. P: Dependent point on posterior wall. C: Cuff point either cervix or vault. Distance to hymen in centimeters (minus above or plus below) after pushing the opposite wall during maximal straining D: Dimensions; base diameter of vestibule/ perineal length.
  The staging system will be interpreted as follows:
  Normal:
  A-3 P-3 C-8 D 2/2
  Stages:
  0: No prolapse.
  A/P-2 OR C-7 to C-2 A,P or C-1 to +1 A,P or C ˃ +1
  X component: (alone or with any stage):
  Dimension disruption: ˃2 or <2

SUMMARY:
There is a strong need for a better, simplified and informative applicable classification system that should be used to speak a common descriptive language among health care providers that treat POP.

The aim of our study is to test our proposed system, assess its validity and value in comparison to the widely used current system (POP-Q).

DETAILED DESCRIPTION:
All patients presented with organ prolapse in the outpatient clinic will be reviewed. Patients are eligible for enrollment in the study when they are complied with all general inclusion criteria, and when none of the exclusion criteria are met after getting written consent from the patients. Study location: (Please provide where the study will be conducted and from where study participants will be recruited) Obstetrics and Gynecology Department, Cairo University Hospital ( Kasr Al Aini), Faculty of Medicine, Cairo University.

All eligible patients will undergo a baseline clinical examination to collect clinical data. This consisted of detailed medical history (including age, parity, detailed obstetric history in the mode of delivery and circumstances associated with each delivery), symptoms, exacerbating and relieving factors, associated symptoms, medication record, history of any previous treatment as pelvic floor muscle training or surgeries, physical examination including weight & height, abdominal and pelvic examination , and clinical category of prolapse according to the POP Q classification system.

Interventions details:

A FIXED APCD classification system will be used to grade the patient symptoms as follows:

A: Associated symptoms:

Incontinence Urgency Constipation Vaginal keratosis/ ulceration

FIXED: the following symptoms will be noted down and graded from 0-10 according to severity:

F: frequency I: infection X: sex problems E: everted mass(external protrusion of mass from the valva as PV lump sensation ,heaviness,itching and ulceration) D: digitation(patient need to digitate to complete the act of micturation or defecation)

APCD: The recruited subject will be examined in lithotomy position. Inspection of the perineum and introitus to look for any vaginal keratosis and measure the introitus length. Examination will be done using sims speculum while the patient is in sims position. The following points will be assessed and noted down as follows:

A: Dependent point on anterior wall. P: Dependent point on posterior wall. C: Cuff point either cervix or vault. Distance to hymen in centimeters (minus above or plus below) after pushing the opposite wall during maximal straining D: Dimensions; base diameter of vestibule/ perineal length.

The staging system will be interpreted as follows:

Normal:

A-3 P-3 C-8 D 2/2

Stages:

0: No prolapse.

1. A/P-2 OR C-7 to C-2
2. A,P or C-1 to +1
3. A,P or C ˃ +1

X component: (alone or with any stage):

Dimension disruption: ˃2 or <2

In order to test the interobserver reliability of the classification system, both history taking and examination will be done by trainee and specialist. The intraobserver reliability will be assessed by repeating the examination by the same examiner two weeks later.

The reliability of the scoring system will be assessed by comparing it to the POP Q classification system, results obtained for each patient at recruitment regarding accuracy and time consumed in the assessed scoring system (using a stopwatch to calculate the time needed for each system applied).

ELIGIBILITY:
Inclusion Criteria:

Age : 18 years and more Symptoms : Pelvic heaviness, urinary symptoms as: stress urinary incontinence, voiding difficulties, dysuria frequency, bowel symptoms as difficulty in defecation sexual symptoms Informed consent

Exclusion Criteria:

Refusal intolerance to the physical examination

* presence of pelvic floor disorders secondary to neurological disease malignancy.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients presented with organ prolapse in the outpatient clinic will be reviewed. Patients were eligible for enrollment in the study when they complied with all general inclusion criteria, and when none of the exclusion criteria were met. After verification of the inclusion and exclusion criteria, written informed consent for the collection of personal medical data was obtained for each patient before enrollment in the study The location of the study will be at theObstetrics and Gynecology Department, Cairo University Hospital ( Kasr Al Aini), Faculty of Medicine, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Inter-observer reliability and validity of the new POP scoring system | one year
  The staging system will be interpreted as follows:
  Normal:
  A-3 P-3 C-8 D 2/2
  Stages:
  0: No prolapse.
  1. A/P-2 OR C-7 to C-2
  2. A,P or C-1 to +1
  3. A,P or C ˃ +1
  X component: (alone or with any stage):
  Dimension disruption: ˃2 or <2

SECONDARY OUTCOMES:
Time required to complete the new classification system | one year
  Time required to complete the new classification system

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf El-Daly, MD, Study Director — Cairo University
Locations (1):
- Doaa Adel, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vergeldt TF, Weemhoff M, IntHout J, Kluivers KB. Risk factors for pelvic organ prolapse and its recurrence: a systematic review. Int Urogynecol J. 2015 Nov;26(11):1559-73. doi: 10.1007/s00192-015-2695-8. Epub 2015 May 13. PMID 25966804
- [Background] Macmillan AK, Merrie AE, Marshall RJ, Parry BR. The prevalence of fecal incontinence in community-dwelling adults: a systematic review of the literature. Dis Colon Rectum. 2004 Aug;47(8):1341-9. doi: 10.1007/s10350-004-0593-0. PMID 15484348
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Kepenekci I, Keskinkilic B, Akinsu F, Cakir P, Elhan AH, Erkek AB, Kuzu MA. Prevalence of pelvic floor disorders in the female population and the impact of age, mode of delivery, and parity. Dis Colon Rectum. 2011 Jan;54(1):85-94. doi: 10.1007/DCR.0b013e3181fd2356. PMID 21160318
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Swift S, Morris S, McKinnie V, Freeman R, Petri E, Scotti RJ, Dwyer P. Validation of a simplified technique for using the POPQ pelvic organ prolapse classification system. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Nov;17(6):615-20. doi: 10.1007/s00192-006-0076-z. Epub 2006 Apr 6. PMID 16598414
- [Background] Lemos N, Korte JE, Iskander M, Freeman R, Arunkalaivanan A, Rizk D, Halaska M, Medina C, Conceicao JC, Parekh M, Martan A, Sorinola O, Wlazlak E, Ghoniem G, Swift S. Center-by-center results of a multicenter prospective trial to determine the inter-observer correlation of the simplified POP-Q in describing pelvic organ prolapse. Int Urogynecol J. 2012 May;23(5):579-84. doi: 10.1007/s00192-011-1593-y. Epub 2011 Nov 15. PMID 22083515
- [Background] Weber AM, Abrams P, Brubaker L, Cundiff G, Davis G, Dmochowski RR, Fischer J, Hull T, Nygaard I, Weidner AC. The standardization of terminology for researchers in female pelvic floor disorders. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(3):178-86. doi: 10.1007/pl00004033. PMID 11451006
- [Background] Slieker-ten Hove MC, Pool-Goudzwaard AL, Eijkemans MJ, Steegers-Theunissen RP, Burger CW, Vierhout ME. Symptomatic pelvic organ prolapse and possible risk factors in a general population. Am J Obstet Gynecol. 2009 Feb;200(2):184.e1-7. doi: 10.1016/j.ajog.2008.08.070. Epub 2008 Dec 25. PMID 19110218
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19110218/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11451006/